CLINICAL TRIAL: NCT01449539
Title: Pilot Study of Hyperbaric Oxygen Therapy in Addition to Standard Growth Factor Support for Hematopoietic Progenitor/Stem Cell Mobilization
Brief Title: Study of Hyperbaric Oxygen Therapy in Addition to Standard Growth Factor Support for Hematopoietic Progenitor/Stem Cell Mobilization
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was terminated early because the site that administered the hyperbaric oxygen treatment closed and an alternative site could not be identified.
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UARK 2010-43
Record Dates: First submitted 2011-09-06; First posted 2011-10-10 (Estimated); Results first posted 2015-02-23 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Multiple Myeloma
Keywords: Hyperbaric oxygen; mobilize; stem cells; growth factor
MeSH Terms: conditions — Multiple Myeloma | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Hyperbaric Oxygen Therapy — Treatment Monday through Friday in a monoplace hyoerbaric chamber 100% oxygen at 2.0 atmospheres (14.7 PSI or the equivalent of being under 33 feet of sea water) for 90 minutes at pressure. Treatment lasts 2 hours as time is allowed for gradual pressurization and depressurization. Each subject will be treated for two weeks for a total of 10 HBOT treatments
  Other Names: HBOT

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of hyperbaric oxygen therapy (HBOT) as a therapeutic option in mobilizing stem cells for autologous stem cell transplant.

DETAILED DESCRIPTION:
Subjects will receive HBOT daily for 10 days in conjunction with standard growth factor treatment regimens for stem cell mobilization. The role of HBOT in stem cell mobilization as well as its role on oxidative stress will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are being considered for autologous stem cell transplant as part of their routine care who have failed at least one prior attempt at stem cell mobilization with any of currently available standard regimens using growth factors.
* Patients in who the use of Mozobil® is medically justified but is not possible because of insurance or financial reasons
* Patients scheduled to begin standard growth factor treatment with Neupogen® as part of routine care.
* Patients who have had a bone marrow evaluation performed within one month prior to enrollment as part of routine clinical care or under IRB# 02815.
* Patients who have had a chest x-ray or CT Chest within 60 days prior to enrollment.
* ECOG performance status ≤ 3 performed within 60 days prior to enrollment which will be determined by history.
* Patients who are at least 18 years of age at the time of registration.
* Patient must have signed an IRB-approved informed consent and understand the investigational nature of the study.

Exclusion Criteria:

* Clinically significant hepatic dysfunction as noted by direct bilirubin or AST >3 times the upper normal limit or clinically significant concurrent hepatitis within 60 days prior to enrollment.
* History of New York Heart Association (NYHA) Class III or Class IV heart failure
* Recent (< 6 months) myocardial infarction, unstable angina, difficult to control congestive heart failure, uncontrolled hypertension, or difficult to control cardiac arrhythmias from medical history.
* Untreated pneumothorax from medical history.
* Uncontrolled seizure disorder from medical history
* Uncontrolled insulin dependent diabetes (verified by routine labs in medical record)
* History of severe claustrophobia
* Severe COPD (FEV1 < 50% of predicted on pulmonary function test) performed within 60 days prior to enrollment
* Untreated ear barotraumas from medical history
* Pregnancy or currently breastfeeding (females of childbearing potential must agree to use adequate contraception during the study). A urine pregnancy test will be performed prior to initiating HBOT.
* Patients currently receiving Bleomycin, Cisplatin, Disulfiram, Doxorubicin, and Sulfamylon.
* Any other condition that the PI determines may jeopardize the safety of the subject during the course of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Waheed, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Science, Little Rock, Arkansas, United States

REFERENCES:
- See also: Related Info — http://www.myeloma.uams.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Hyperbaric Oxygen Therapy: Daily HBOT treatments (100% oxygen at 2.0 atmospheres (14.7) PSI for 90 minutes) for 10 days (Monday-Friday for two weeks) in conjunction with standard growth factor treatment regimens
Period: Overall Study
Arm/Group | Hyperbaric Oxygen Therapy
Started | 8
Completed | 4
Not Completed | 4
Not completed — Withdrawal by Subject | 3
Not completed — Toxicity not study related | 1

BASELINE CHARACTERISTICS:
Groups:
- Hyperbaric Oxygen Therapy: Treatment Monday through Friday in a monoplace hyperbaric chamber 100% oxygen at 2.0 atmospheres for 90 minutes at pressure. Treatment lasts about 2 hours as time is allowed for gradual pressurization and depressurization. Treated for two weeks a total of 10 HBOT treatments.
Arm/Group | Hyperbaric Oxygen Therapy
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.25 (50.185)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Stem Cells Collected
Description: Total stem cells collected from all participants at one week post-study treatment
Time Frame: one week post-treatment
Population: Four of eight enrolled subjects completed the study.
Measure: Number; unit: stem cells
Groups:
- Hyperbaric Oxygen Therapy: Treatment Monday through Friday in a monoplace hyperbaric chamber 100% oxygen at 2.0 atmospheres (the equivalent of being under 33 feet of sea water) for 90 minutes. Treatment lasts 2 hours as time is allowed for gradual pressurization and depressurization. Each participant will be treated for two weeks for a total of 10 HBOT treatments.
Arm/Group | Hyperbaric Oxygen Therapy
Number analyzed (Participants) | 4
stem cells | 8910000

ADVERSE EVENTS:
Time Frame: Approximately 6 months.
Arm/Group | Hyperbaric Oxygen Therapy
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 8/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hyperbaric Oxygen Therapy (N=8)
ALP Increased (Blood and lymphatic system disorders) | 5
Alopecia (General disorders) | 1
Anemia (Blood and lymphatic system disorders) | 8
Auditory/Ear-other (Ear and labyrinth disorders) | 1
Bicarbonate decrease (Blood and lymphatic system disorders) | 3
Bruising (Skin and subcutaneous tissue disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Creatinine Increased (Metabolism and nutrition disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Fatigue (General disorders) | 3
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 8
Hypoalbuminemia (Blood and lymphatic system disorders) | 8
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 4
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Upper airway - NOS (Respiratory, thoracic and mediastinal disorders) | 1
Pain - Buttock (General disorders) | 1
Pain - Middle ear (Ear and labyrinth disorders) | 2
Pain - upper back (General disorders) | 1
Pain - joint (General disorders) | 1
Pulmonary - other (Respiratory, thoracic and mediastinal disorders) | 1
SGOT Increased (Blood and lymphatic system disorders) | 1
SGPT Increased (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 8
Leukopenia (Blood and lymphatic system disorders) | 4

LIMITATIONS AND CAVEATS:
Study was terminated early because the site that administered the hyperbaric oxygen treatment closed and an alternative site could not be identified. Only four subjects completed the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No